CLINICAL TRIAL: NCT05077488
Title: Prospective, Open Label, Study to Evaluate VOLIFT With Lidocaine Treatment for FORehead Contouring and Marionette Lines
Brief Title: VFORM: Prospective, Open Label, Study to Evaluate VOLIFT With Lidocaine Treatment for FORehead Contouring and Marionette Lines
Acronym: VFORM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Collaborators: Eurofins Dermscan Pharmascan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED-MA-FAS-0651; 2021-A00606-35 (Other: ANSM)
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Marionette Lines Forehead Contouring
Keywords: skin depressions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Juvéderm® VOLIFT™ with Lidocaine (Experimental): Intradermal injection (deep dermis) in marionettes lines and/or forehead by a specialist injector
  Interventions: Device: Juvéderm® VOLIFT™ with Lidocaine

INTERVENTIONS:
Device: Juvéderm® VOLIFT™ with Lidocaine — Sterile gel in disposable syringe

SUMMARY:
To collect post-marketing data on Juvéderm® VOLIFT™ with Lidocaine on the following indications:

1. Marionette lines (treatment skin depressions)
2. Forehead contouring (face contouring)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age or older.
2. Signed the Independent Ethics Committee (IEC)-approved informed consent form prior to any studyrelated procedures being performed.
3. Eligible for treatment in at least one of the following treatment areas:

   1. Juvéderm VOLIFT treatment of skin depressions in the marionette lines:

      * Grade 1, 2, 3 or 4 on both sides at baseline in the Allergan Marionette Line Scale
      * Juvéderm VOLIFT is permitted in the oral commissures, at the discretion of the subject and investigator
   2. Juvéderm VOLIFT treatment for irregularities of forehead contouring as assessed by the investigator and is likely to see improvement
4. Accept the obligation not to receive any other facial procedures or treatments anywhere in the face during the study that are not related to the study.
5. Women of childbearing potential must have a negative urine pregnancy test before each injectable treatment and practice a reliable method of contraception throughout the study.
6. Ability to follow study instructions and likely to complete all required visits and assessments, as assessed by the Investigator.
7. Affiliated to a health social security system.

Exclusion Criteria:

In terms of population

1. Females who are pregnant, nursing, or planning a pregnancy.
2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
3. Subject in a social or sanitary establishment (socially or mentally vulnerable).
4. Current enrolment in an investigational drug or device study, participation in such a study within 6 weeks before enrollment, or be planning to participate in another investigation during the course of this study.
5. Is an employee (or immediate relative of an employee) of the Investigator, study staff, Allergan, or a representative of Allergan.
6. In France: subject having received 4500 euros indemnities for participation in researches involving human beings in the 12 previous months, including participation in the present study.

   In terms of associated pathology
7. Has a history of multiple or severe allergies, anaphylaxis, atopy, or allergy to lidocaine, HA products, or Streptococcal protein, or is planning to undergo desensitization therapy during the study.
8. Has an active inflammation or infection (acne, herpes,…), cancerous or precancerous lesion, or unhealed wound.
9. Subject with history of hypertrophic scarring
10. Has porphyria.
11. Has epilepsy.
12. Has impaired cardiac conduction, severely impaired hepatic function, or severe renal dysfunction.
13. History of, or currently suffering from, autoimmune disease or autoimmune deficiency or being under immunosuppressive therapy.
14. History of streptococcal disease (recurrent sore throats, acute rheumatic fever).
15. Has any uncontrolled disease.
16. Has any condition or is in a situation that, in the Investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study. Relating to previous or ongoing treatment
17. Has ever undergone facial plastic surgery or received permanent facial implants (e.g., polymethylmethacrylate, silicone, polytetrafluoroethylene, threads) anywhere in the face, or is planning to be implanted with any of these products during the study.
18. Has undergone semi-permanent dermal filler treatment (e.g., hyaluronic acid, calcium hydroxyapatite, poly-L-lactic acid) in the face within 12 months before enrolment or is planning to undergo such treatment during the study.
19. Has undergone mesotherapy or cosmetic resurfacing (laser, photo-modulation, intense pulsed light, radiofrequency, dermabrasion, chemical peel, or other ablative or non-ablative procedures) anywhere in the face or neck, or Botulinum toxin injections in the face within 6 months before enrolment or is planning to undergo any of these procedures during the study.
20. Has begun using any over-the-counter or prescription, oral or topical, anti-wrinkle products within 90 days before enrolment or is planning to begin using such products during the study (subjects who have been on a regimen of such products for at least 90 days are eligible for the study if they intend to continue their regimen throughout the study).
21. Is on an ongoing regimen of anti-coagulation therapy (e.g., warfarin) or non-steroidal antiinflammatory drugs (NSAIDs) (e.g., aspirin, ibuprofen) or other substances known to increase coagulation time (e.g., herbal supplements with garlic or gingko) within 10 days of undergoing study device treatment (study treatment may be delayed as necessary to accommodate this 10- day washout period).
22. Is on a concurrent regimen of lidocaine or structurally related local anaesthetics (e.g., bupivacaine).
23. Is on an ongoing treatment that reduce or inhibit hepatic metabolism (cimetidine, beta-blockers, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Forehead Contouring: Proportion of subjects with a Global Aesthetic Improvement Scale (GAIS) equal to 'improved" or "much improved" as assessed by a blinded aesthetic doctor of the contouring of the forehead using a 3D image. | Baseline to 30 Days
  The Global Aesthetic Improvement Scale is a 5-point scale ranging from "Much Improved" to "Much Worse" and it is used for the assessment of the level of improvement to the subjects forehead contouring
Marionette Lines: Proportion of subjects with a ≥1-point change in the Marionette Line scale from baseline before treatment to 30 days post treatment. | Baseline to 30 Days
  The Marionette Line scale is a 5-point scale ranging from 0 (None- No Lines) to 4 (Very Severe) and it is used for the assessment of the level of improvement to the subjects marionette lines

SECONDARY OUTCOMES:
Forehead Contouring: Change in overall FACE-Q Satisfaction with Facial Appearance score from baseline to 30 days, 3 months, 6 months, 9 months, 12 months | Baseline to 30 days, 3 months, 6 months, 9 months, 12 months
  The FACE-Q™ is a validated 10 question assessment measuring how satisfied the participant is with their facial appearance. Each question is answered on a 4-point scale where: 1=Very Dissatisfied, 2=Somewhat dissatisfied, 3=Somewhat satisfied, and 4= Very Satisfied. The responses to the items were converted to a 100-point Rausch transformed scale score: 0 (worst) to 100 (best). Higher scores indicate higher satisfaction. A positive change from Baseline indicates improvement.
Marionette Lines: Proportion of subjects with a ≥1-point change in the Allergan Marionette Line scale from baseline before treatment to 3 months, 6 months, 9 months, 12 months | Baseline before treatment to 3 months, 6 months, 9 months, 12 months
  The Marionette Line scale is a 5-point scale ranging from 0 (None- No Lines) to 4 (Very Severe) and it is used for the assessment of the level of improvement to the subjects marionette lines
Forehead Contouring: Proportion of subjects with a GAIS equal to 'improved" or "much improved" as assessed by a blinded aesthetic doctor using a 3D image at 3 months, 6 months, 9 months and 12 months | 3 months, 6 months, 9 months and 12 months
  The Global Aesthetic Improvement Scale is a 5-point scale ranging from "Much Improved" to "Much Worse" and it is used for the assessment of the level of improvement to the subjects forehead contouring
Marionette Lines: Change in overall FACE-Q Satisfaction with Facial Appearance score from baseline to 30 days, 3 months, 6 months, 9 months, 12 months | Baseline to 12 Months
  The FACE-Q™ is a validated 10 question assessment measuring how satisfied the participant is with their facial appearance. Each question is answered on a 4-point scale where: 1=Very Dissatisfied, 2=Somewhat dissatisfied, 3=Somewhat satisfied, and 4= Very Satisfied. The responses to the items were converted to a 100-point Rausch transformed scale score: 0 (worst) to 100 (best). Higher scores indicate higher satisfaction. A positive change from Baseline indicates improvement.
Forehead Contouring: Proportion of subjects with a GAIS equal to 'improved" or "much improved" as assessed by the investigator using baseline 2D photographs (live evaluation) at 30 days, 3 months, 6 months, 9 months and 12 months | 30 days to 12 Months
  The Global Aesthetic Improvement Scale is a 5-point scale ranging from "Much Improved" to "Much Worse" and it is used for the assessment of the level of improvement to the subjects forehead contouring
Marionette Lines: Change in overall FACE-Q Appraisal of lines: marionette score from baseline to all administered timepoints | Baseline to 12 Months
  The participant assessed appraisal of marionette lines using the FACE-Q questionnaire measured on a 4-point scale where 1=Not At All, 2=A Little, 3=Moderately , 4=Extremely. The responses to the items on the questionnaire are converted to a 100-point Rasch transformed scale score with 0 (worst) to 100 (best). A positive change from Baseline indicates improvement.
Forehead Contouring: Proportion of subjects with a GAIS equal to 'improved" or "much improved" as assessed by the subjects using baseline 2D photographs (live evaluation) at 30 days, 3 months, 6 months, 9 months and 12 months | 30 days, 3 months, 6 months, 9 months and 12 months
  The Global Aesthetic Improvement Scale is a 5-point scale ranging from "Much Improved" to "Much Worse" and it is used for the assessment of the level of improvement to the subjects forehead contouring
Marionette Lines: Proportion of subjects with a GAIS equal to 'improved" or "much improved" as assessed by the investigator using baseline 2D photographs (live evaluation) at 30 days, 3 months, 6 months, 9 months and 12 months | 30 days, 3 months, 6 months, 9 months and 12 months
  The Global Aesthetic Improvement Scale is a 5-point scale ranging from "Much Improved" to "Much Worse" and it is used for the assessment of the level of improvement to the subjects marionette lines
Forehead Contouring: Volume change in the forehead using 3D imaging from baseline before treatment to 30 days, 3 months, 6 months, 9 months, 12 months | 30 days, 3 months, 6 months, 9 months, 12 months
Marionette Lines: Volume change in the marionette lines using 3D imaging from baseline before treatment to 30 days, 3 months, 6 months, 9 months, 12 months | 30 days, 3 months, 6 months, 9 months, 12 months
Forehead Contouring: Contour changes in the forehead using 3D imaging from baseline before treatment to 30 days, 3 months, 6 months, 9 months, 12 months | 30 days, 3 months, 6 months, 9 months, 12 months
Marionette Lines: Proportion of subjects with a GAIS equal to 'improved" or "much improved" as assessed by the subjects using baseline 2D photographs (live evaluation) at 30 days, 3 months, 6 months, 9 months and 12 months | 30 days, 3 months, 6 months, 9 months and 12 months
  The Global Aesthetic Improvement Scale is a 5-point scale ranging from "Much Improved" to "Much Worse" and it is used for the assessment of the level of improvement to the subjects marionette lines

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (1):
- Eurofins Pharmascan /ID# 243454, Lyon, France

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/